CLINICAL TRIAL: NCT06510114
Title: Comparison of Two Intravenous Methylprednisolone Protocols in Patients With Graves Orbitopathy: a Randomized Clinical Trial
Brief Title: A Randomized Clinical Trial of Intravenous Methylprednisolone With 2 Protocols in Patients With Graves Orbitopathy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shuo Lin, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG2024-016-01
Record Dates: First submitted 2024-06-24; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Graves Ophthalmopathy
Keywords: Hyperthyroidism; Graves Ophthalmopathy; glucocorticoid
MeSH Terms: conditions — Graves Ophthalmopathy; Hyperthyroidism | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Participants with active moderate-to-severe GO were randomized at a ratio of 1:1 to receive glucocorticoid therapy for 12 weeks on a weekly protocol or daily scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The daily scheme was as follows: 0.5 g methylprednisolone i.v. daily for 5 consecutive days, followed by oral prednisone for 6 months. Oral prednisone started at 40 mg/day for 4 weeks and then the dose was tapered by 5 mg/day every 2-4 weeks.
  Interventions: Drug: methylprednisolone(daily scheme)
- Group B (Active Comparator): The weekly protocol was as follows: 0.5 g methylprednisolone i.v. weekly for 6 weeks and then the dose was tapered by 0.25 g/week over the following 6 weeks.
  Interventions: Drug: methylprednisolone(weekly scheme)

INTERVENTIONS:
Drug: methylprednisolone(daily scheme) — 0.5 g methylprednisolone i.v. daily for 5 consecutive days, followed by oral prednisone for 6 months. Oral prednisone started at 40 mg/day for 4 weeks and then the dose was tapered by 5 mg/day every 2-4 weeks.
  Other Names: prednisone
  Arms: Group A
Drug: methylprednisolone(weekly scheme) — 0.5 g methylprednisolone i.v. weekly for 6 weeks and then the dose was tapered by 0.25 g/week over the following 6 weeks.
  Arms: Group B

SUMMARY:
Intravenous glucocorticoid (IVGC) is an accessible and effective therapy for Graves orbitopathy (GO); the 4.5-g weekly protocol is well studied, but many details of treatment protocols need to be clarified. The goal of this trial is to compare the efficacy and safety of weekly and daily protocol of IVGC in GO. Researchers will compare daily protocol to weekly protocol to see if daily protocol works to treat GO.

DETAILED DESCRIPTION:
The goal of this trial is to compare the efficacy and safety of weekly and daily protocol of IVGC in GO.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old;
2. diagnosed as thyroid associated ophthalmopathy by using Bartley criteria，Moderate to severe (EUGOGO grade), with CAS≥3 points;
3. Thyroid function normally lasts for more than 2 months, with oral antithyroid drugs or thyroid surgery, or six months after iodine-131 treatment;
4. without receiving immunosuppressive therapy for thyroid eye disease before.

Exclusion Criteria:

(1) severe cardiac, liver and renal insufficiency (2) acute or chronic viral hepatitis or tuberculosis (3) optic neuropathy (4) received immunosuppressive and glucocorticoid therapy for any reason within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the overall response rate at 24 week | 24 week
  "Response" was defined as an improvement in at least two of the following four criteria were present, and the contralateral eye disease did not worsen: (1) the width of the eyelid was reduced by ≥2 mm; (2) The five scores of eyelid congestion, eyelid edema, conjunctival congestion, conjunctival edema and carunculae lacrimalis swelling in CAS decreased by ≥1 point; (3) The regression of exophthalmos ≥2 mm; (4) Increased eye movement ≥8° or improved diplopia ≥ grade I (continuous to interrupted, interrupted to brief, brief to none).

SECONDARY OUTCOMES:
Changes of clinical activity score (CAS) from baseline to 24 week | 24 week
  changes of clinical activity score (CAS) from baseline to 24 week
changes of quality of life score (QoF-s) from baseline to 24 week | 24 week
  changes of quality of life score (QoF-s )
changes of exophthalmos from baseline to 24 week | 24 week
  changes of exophthalmos from baseline to 24 week
changes of width of the eyelid from baseline to 24 week | 24 week
  changes of width of the eyelid from baseline to 24 week
changes of diplopia grade from baseline to 24 week | 24 week
  changes of diplopia grade from baseline to 24 week

OTHER OUTCOMES:
Changes of blood pressure from baseline to 24 week | 24 week
  Changes of blood pressure from baseline to 24 week
Changes of weight from baseline to 24 week | 24 week
  Changes of weight from baseline to 24 week
Changes of fasting blood glucose from baseline to 24 week | 24 week
  Changes of fasting blood glucose from baseline to 24 week
Changes of serum low density lipoprotein cholesterol | 24 week
  Changes of low density lipoprotein cholesterol from baseline to 24 week
Changes of serum triglyceride | 24 week
  Changes of serum triglyceride from baseline to 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Lin, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No